CLINICAL TRIAL: NCT00987831
Title: Biomarkers of Lupus Disease: Study of Biomarker Changes Before and After Treatment With Depomedrol and Background Medication Withdrawal in Patients With Mild to Moderate SLE Disease Activity
Brief Title: Biomarkers of Lupus Disease: Serial Biomarker Sampling in Patients With Active Systemic Lupus Erythematosus (SLE)
Acronym: BOLD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Joan Merrill, MD, Head, Clinical Pharmacology Research Program, Oklahoma Medical Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMRF 09-02; Pfizer Inc (Other Grant/Funding Number: Pfizer investigator initiated study)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; lupus; biomarkers; depomedrol; flare; disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Blood drawing only Group C (Experimental): Healthy controls, age, sex and ethnicity matched to the active study participants were recruited for two time blood donation as controls for the biomarker studies
  Interventions: Other: Blood drawing only Group C
- Group A SLE prospective study (Experimental): In Group A SLE patients enter with active disease. Any immune suppressant (e.g. methotrexate, azathioprine or mmf) is withdrawn and after blood drawing, depomedrol up to 160 mg IM is given. This may be repeated for a maximum of 160mg up to four times total in the first two weeks. Depomedrol is expected to last 1-3 months, serial biomarkers will be drawn until time of flare, at which time biomarkers will be drawn, patient is defined as meeting endpoint and new treatment initiated. Patients may elect to continue to donate blood samples per protocol up to one year.
  Interventions: Drug: Group A SLE prospective study
- Group B SLE one blood donation (Experimental): SLE patients who meet the same entry criteria as Group A could elect to donate blood one time and not to continue in the prospective protocol. No extra intervention was performed other than blood draw and medical records review. This allowed an extension of cross sectional comparisons between biomarker changes related to background treatments by combining Group A baseline data with Group B data.
  Interventions: Other: Group B SLE one blood donation

INTERVENTIONS:
Other: Group B SLE one blood donation — Blood drawing, history, physical examination,medical record review, questionnaires, completion of disease activity measures including SLEDAI,BILAG, CLASI,PGA,PROs,LFA investigational systems, BICLA, SRI
  Arms: Group B SLE one blood donation
Other: Blood drawing only Group C — Blood drawing and Brief medical history to ensure status of healthy control
  Arms: Blood drawing only Group C
Drug: Group A SLE prospective study — Patients have history and physical exmamination at each visit. Blood is drawn at each visit. At baseline, any background immune suppressant is stopped and patients given depomedrol up to 160 mg IM which can be repeated up to four times in the first two weeks. Patients are seen again at week 2, 4 and monthly until the final flare visit at which time they donate blood, receive appropriate treatments and exit study. Patients may elect to continue in study for up to one year. The following disease activity measures are included: SLEDAI, BILAG, CLASI, PGA, PROs (including lupus PRO and SF-36 ant ptGA), joint counts, exploratory outcome measures,BICLA,SRI
  Other Names: depomedrol; medrol; methylprednisolone
  Arms: Group A SLE prospective study

SUMMARY:
Hypothesis: A reason for repeated disappointing outcomes of clinical trials testing targeted immune biologics for lupus may be the heterogeneity of the disease, exacerbated by the variable effects on immune homeostasis of the background medications that must be continued, in most study designs, in these flare-prone patients.

Purpose of Study: This study was designed to purposefully study a population equivalent to the placebo group of typical trials in SLE. In Group A patients entered the trial in mild-moderate flare, were treated with depomedrol, and any background immune suppressants withdrawn. Biomarkers at entry on various medications can be compared to biomarkers after steroid efficacy with background immune suppressants withdrawn. Depomedrol usually wears off over one to three months. Patients were closely observed, with serial biomarkers drawn at monthly intervals or immediately at the time of a new flare. Those patients developing new flares donated blood samples, were immediately treated as deemed appropriate, exiting the study. Group A was designed for up to 50 patients and recruited a total of 41. An additional group of 62 SLE patients donated blood once without additional interventions in order to increase the power of exploratory cross-sectional biomarker analysis on different immune suppressants (Group B). A control population of matched, healthy individuals donated blood twice for the same biomarker studies to validate these assays (Group C).

DETAILED DESCRIPTION:
Original Protocol for Group A: Patients with at least a SLEDAI score of 6 or a BILAG score of B in at least two organ systems or A in at least one organ system were immediately entered into this study once informed consent was obtained. Background immune suppressants (if any) were stopped and in about half of the patients hydroxychloroquine was also stopped. All patients immediately received a shot of depomedrol 160 mg IM. Over the next two weeks they could elect up to three more shots of depomedrol for a total of four shots by the two week visit period. A complete battery of blood tests to assess lupus disease was drawn at the screening visit, and monthly thereafter. Exploratory biomarker studies were drawn as often as weekly for some markers and as often as three times in the study (landmark visits) for others. Protocol Changes during course of study: Biomarkers were drawn at Day zero, week 2 week 4 and monthly thereafter until flare. Patients who did not improve with protocol steroid treatments were withdrawn from Group A and immediately treated as warranted. Since there was no protocol-defined improving visit, they could not continue the protocol until flare. However their baseline samples were appropriate for study as part of Group B (see below).

Landmark visits for Group A are defined as: 1.) screening (pre-dose, on background meds with active disease) 2.) two weeks or four weeks after screening as optimal to assess a patient who has stopped background meds and is now maximally improved (but at least one grade drop in BILAG scores in all organs entered at A or B or a four point drop in SLEDAI, otherwise the participant is deemed a treatment failure and could not participate further in Group A. 3.) Flare visit on no background immune suppression defined as an increase in SLEDAI of 4 points from maximal improvement or one new BILAG moderate (B) score AND the investigator considers the condition to be a significant flare with intent to treat. Patients were (whenever possible) seen within 3 days for the flare visit if flare occured between monthly scheduled visits.

The primary purpose of this study was to evaluate the time to flare and safety of a treatment withdrawal protocol in patients with active, but non-organ threatening SLE. The following biomarkers were obtained for exploratory analysis: cytokine panel, B Cell studies, T Cell studies, autoantibody profiles, epigenetic and gene expression studies and flow cytometry studies.

ELIGIBILITY:
Inclusion Criteria:

SLE Groups (Group A and B):

1. ACR criteria for SLE.
2. At least two organ systems moderately active to a minimum of BILAG B or SLEDAI score of 6.

Control group (Group C):

1. Age, ethnicity and gender matched (2:1) with an SLE study participant.
2. Free of active or major chronic disease as determined by brief history.

Exclusion Criteria:

1. Safety or circumstantial reasons why volunteer cannot comply with the protocol.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan T Merrill, Principal Investigator — Oklahoma Medical Research Foundation
Locations (2):
- United States (2):
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Pfizer Inc, Collegeville, Pennsylvania

REFERENCES:
- [Derived] Merrill JT, Immermann F, Whitley M, Zhou T, Hill A, O'Toole M, Reddy P, Honczarenko M, Thanou A, Rawdon J, Guthridge JM, James JA, Sridharan S. The Biomarkers of Lupus Disease Study: A Bold Approach May Mitigate Interference of Background Immunosuppressants in Clinical Trials. Arthritis Rheumatol. 2017 Jun;69(6):1257-1266. doi: 10.1002/art.40086. PMID 28257602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The final recruitment tally is as follows: 41 SLE patients entered the prospective serial blood donation study. 62 SLE patients gave one time blood sample and 52 controls gave two blood samples each
Pre-assignment Details: All patients in Group A (prospective study) had any immune suppressive (e.g. MMF, MTX, AZA) withdrawn at the time of entry and all received between 1-3 depomedrol shots up to 160 mg each. Those who did not improve were immediately withdrawn from prospective study but the original sample was retained, in all cases, for the cross sectional arm.
Groups:
- Group A Medication Withdrawal, Depomedrol, Prospective Follow-: When depomedrol was given, any immune suppressant being taken (e.g. aza, mmf, mtx) was stopped and biomarkers studied before and after this change. Depomedrol was expected to last 1-3 months, serial biomarkers were drawn until time of any flare, designated as end of study. Patients could elect to continue to donate blood samples per protocol up to one year. Of 41 patients who improved after depomedrol and could complete Group A, 40 flared at or before the six month visit. One patient continued for one year and did not flare. This study design allowed the comparison of 40 patients flaring at baseline on or not on background immune suppression vs themselves serving as their own control flaring later....not on immune suppression.
- Group C Healthy Controls: Healthy controls, age, sex and ethnicity matched to SLE study participants were recruited for two time blood donation as controls for the biomarker studies
  Blood drawing and brief history only : No treatments given
- Group B SLE One Time Donation: We amended protocol with IRB approval to include more patients in this group and ended up recruiting a total of 62. This was to allow enrichment of a cross sectional study of biomarkers related to the different background immune suppressants used in Group A at baseline. By combining baseline samples from Group A and Group B data we had a total of 103 lupus samples to study cross sectionally comparing impact of methotrexate, mmf, azathioprine or no IS on a range of biomarkers.
Period: Overall Study
Arm/Group | Group A Medication Withdrawal, Depomedrol, Prospective Follow- | Group C Healthy Controls | Group B SLE One Time Donation
Started | 41 (41 patients improved after depomedrol, if not improved, treated and moved to Group B) | 55 (52 healthy controls donated biomarkers on two occasions in order to verify biomarkers ranges) | 62 (Anyone who entered this arm completed it the same day)
Completed | 40 (40 patients completed in 6 months. 1 patient did not meet completion definition in 12 months.) | 52 (all controls returned for two visits) | 62 (Anyone who entered this arm completed it the same day)
Not Completed | 1 | 3 | 0
Not completed — Never flared in 12 months | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A Medication Withdrawal, Depomedrol, Prospective Follow-: When depomedrol was given, any immune suppressant being taken (e.g. aza, mmf, mtx) was stopped and biomarkers studied before and after this change. Depomedrol was expected to last 1-3 months, serial biomarkers were drawn until time of any flare, designated as end of study. Patients could elect to continue to donate blood samples per protocol up to one year. Of 41 patients who improved after depomedrol and could complete Group A, 40 flared at or before the six month visit. One patient continued for one year and did not flare. This study design allowed the comparison of 40 patients flaring at baseline on or not on background immune suppresion vs themselves serving as their own control flaring later....not on immune suppression.
- Total: Total of all reporting groups
Arm/Group | Group A Medication Withdrawal, Depomedrol, Prospective Follow- | Group C Healthy Controls | Group B SLE One Time Donation | Total
Number analyzed (Participants) | 41 | 55 | 62 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 55 | 62 | 157
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.9) | 40.8 (12.1) | 41.6 (11.3) | 41.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 53 | 55 | 147
  Male | 2 | 2 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 41 | 55 | 62 | 158

OUTCOME MEASURES:

1. Primary Outcome: Time to Flare Comparing Patients With Moderate vs Severe Disease Activity at Baseline
Description: Group A only: patients on immunosuppressive treatments had them withdrawn at baseline. All patients were allowed up to 160 mg depomedrol at baseline which could be repeated within two weeks up to a total of 4 shots maximum or until satisfactory improvement. Time to flare was calculated from baseline. moderate disease at baseline was defined as up to 3 BILAG B (moderate disease) organ scores, no BILAG A (severe disease) score and a SLEDAI </= 10. Severe disease required >3 BILAG B, OR at least one BILAG A OR SLEDAI > 10 or meeting criteria for a severe flare on the SELENA SLEDAI flare index. At baseline 25 patients with moderate disease. 16 patients had severe disease. Note: severe rash with A on BILAG is only SLEDAI=2, explaining some discrepancies in measures
Time Frame: 12 months
Population: This prespecified primary outcome was restricted to Group A only. This was an exploratory proof of concept study, not powered for the primary endpoint
Measure: Median (95% Confidence Interval); unit: days to flare
Groups:
- Severe Disease Activity at Baseline: This is fully explained above. Severe disease activity is defined as > 3 BILAG B, OR at least one BILAG A or SLEDAI > 10 OR Meets Definition for severe Flare on SELENA SLEDAI
- Moderate Disease Activity at Baseline: this is fully explained above. Moderate disease activity is defined as up to 3 BILAG B, no A, and SLEDAI </= 10.
Arm/Group | Severe Disease Activity at Baseline | Moderate Disease Activity at Baseline
Number analyzed (Participants) | 16 | 25
days to flare | 45 [30 to 91] | 71 [43 to 91]
Statistical Analysis 1: Comparison: Severe Disease Activity at Baseline vs Moderate Disease Activity at Baseline; Test type: Superiority or Other; p = 0.2738, Log Rank — Definition of Moderate Disease was </= 3 BILAG B (moderate) organ scores, no A (severe) scores and SLEDAI </=10. Severe disease was > 3 BILAG B or >/= BILAG A or SLEDAI > 10 or meets definition for severe flare on the SELENA SLEDAI Flare Index; Median Difference (Final Values) = 30, 95% CI 2-sided [5 to 95]

2. Post Hoc Outcome: Time to Flare Comparing Patients With (at Baseline) British Isles Lupus Assessment Group Index (BILAG) >/= 17 (Severe Disease) to Those With BILAG < 17 (Moderate Disease Activity).
Time Frame: 12 months
Population: Only 40/41 entered patients completed the study by the definition of the endpoint which was flare.
Measure: Median (95% Confidence Interval); unit: days to flare
Groups:
- Severe Disease Activity at Baseline: This is fully explained above. Severe disease is now defined as total cumulative BILAG score >/= 17
- Moderate Disease Activity at Baseline: this is fully explained above. Moderate disease is now defined as BILAG < 17 in cumulative score
Arm/Group | Severe Disease Activity at Baseline | Moderate Disease Activity at Baseline
Number analyzed (Participants) | 11 | 29
days to flare | 40 [29 to 72] | 72.5 [46 to 99]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until end of study participation (ranging one visit to 12 months) Note all patients in Group A who flared were treated and followed up within six weeks and all improved again on new treatments initiated at the time of flare.
Description: This was an interventional study using depomedrol which is a commonly used treatment in our clinic. The main safety issue in the study was the withdrawal of background immune suppressants.
Arm/Group | Group A Medication Withdrawal, Depomedrol, Prospective Follow- | Group C Healthy Controls | Group B SLE One Time Donation
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/55 | 0/62
Other Adverse Events (participants affected / at risk) | 29/41 | 0/55 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Medication Withdrawal, Depomedrol, Prospective Follow- (N=41) | Group C Healthy Controls (N=55) | Group B SLE One Time Donation (N=62)
Bleeding Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — The patient developed severe abdominal pain and was hospitalized for four days. Found to have an actively bleeding peptic ulcer. She recovered completely with supportive care and medications.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A Medication Withdrawal, Depomedrol, Prospective Follow- (N=41) | Group C Healthy Controls (N=55) | Group B SLE One Time Donation (N=62)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) — 3 total upper respiratory infections reported. Maximum severity was moderate. All resolved without sequelae.
sinusitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) — 4 reports of sinusitis. Maximum severity was moderate. All resolved without sequelae.
urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) — There were 2 reports of UTI. Both resolved without sequelae.
gastroenteritis (Gastrointestinal disorders) | 8 (8) | 0 (0) | 0 (0) — There were eight reports of abdominal discomfort, abdominal distress, non specific abdominal pains only one of which was later found to be in a patient positive for H pylori. All conditions improved without sequelae
oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) — 2 cases of oral candidiasis which may have been related to steroid therapy in protocol. Both resolved with treatment
cushingoid face (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) — 2 reports of cushinoid face which could be related to steroid therapy in study. However other steroids had been used.
insomnia (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) — 4 reports of insomnia which could be related to steroid therapy in protocol. None were clinically significant
seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) — two reports of seasonal allergies which would be expected in these patients
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — reports of back and hip pain, non specific, unlikely to be due to lupus or the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less